CLINICAL TRIAL: NCT00304746
Title: A Parallel-Group, Placebo-Controlled Trial of AndroGel in Men With Major Depressive Disorder Who Display an Incomplete Response to Standard Antidepressant Treatment
Brief Title: AndroGel in Men With Major Depression and Incomplete Response to Antidepressant Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: Solvay Pharmaceuticals (Industry)
Responsible Party: Harrison G. Pope, Jr., M.D., McLean Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2005P-001667
Record Dates: First submitted 2006-03-16; First posted 2006-03-20 (Estimated); Results first posted 2010-11-17 (Estimated); Last update posted 2010-11-24 (Estimated); Status verified 2010-11

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Testosterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- testosterone gel (Active Comparator): AndroGel (1% testosterone transdermal gel), 2.5 g to 10 g daily
  Interventions: Drug: Testosterone gel
- placebo gel (Placebo Comparator): Placebo gel
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Testosterone gel — AndroGel 2.5g and 5g sachets at doses ranging from 10g/day for duration of trial.
  Other Names: AndroGel
  Arms: testosterone gel
Drug: Placebo — Placebo
  Arms: placebo gel

SUMMARY:
We hypothesize that AndroGel may offer some relief to subjects with low or borderline testosterone levels who suffer from depression and have failed to respond to a trial of a standard antidepressant.

During this nine week, outpatient, double-blind study, male subjects between the ages of 30 and 65 years with treatment-refractory depression and low or borderline low testosterone levels will be treated with either AndroGel or placebo. Following this nine week, double-blind phase, eligible subjects will have the option to continue into a six month, open-label phase during which time all subjects will receive the AndroGel patch.

DETAILED DESCRIPTION:
We will recruit 100 men between the ages of 30 and 65 years who have treatment-refractory depression and low or borderline low testosterone levels for participation in this study. For a period of nine weeks subjects will receive double-blind treatment with either AndroGel (testosterone gel) or placebo. During this double-blind treatment phase subjects will come to McLean Hospital for a total of seven visits. Both clinical assessments (including ratings of your levels of depression and anxiety, quality of life, and visuospatial memory)and laboratory tests will be performed at these visits. Following the nine week, double-blind phase, eligible subjects may enter into a six month, open-label treatment phase in which all subject receive AndroGel. If you participate in the open-label phase, you will be asked to return to the site for 8 visits during the six month period.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 30-65 years old
* Taking at least one serotonergic antidepressant at adequate dose for at least six weeks but still meeting DSM-IV criteria for major depressive disorder within the past year
* HAM-D score >12

Exclusion Criteria:

* Current suicidal ideation
* Substance abuse or dependence within the past year
* Current or past psychotic symptoms
* A history of bipolar disorder
* A prostate-specific antigen (PSA) level greater than 4.0 ng/ml
* Other clinically significant medical condition
* A history of failing to show any clinically significant response to two or more adequate trials of different antidepressants.

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2006-04; Primary Completion 2008-12 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harrison G Pope, M.D., Principal Investigator — Mclean Hospital; Stuart N Seidman, M.D., Principal Investigator — Columbia University
Locations (2):
- McLean Hospital, Belmont, Massachusetts, United States
- The Chaim Sheba Medical Center, Tel Litwinsky, Israel

REFERENCES:
- [Result] Pope HG Jr, Amiaz R, Brennan BP, Orr G, Weiser M, Kelly JF, Kanayama G, Siegel A, Hudson JI, Seidman SN. Parallel-group placebo-controlled trial of testosterone gel in men with major depressive disorder displaying an incomplete response to standard antidepressant treatment. J Clin Psychopharmacol. 2010 Apr;30(2):126-34. doi: 10.1097/JCP.0b013e3181d207ca. PMID 20520285

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at two sites - McLean Hospital in Belmont Massachusetts, USA and the Chaim Sheba Medical Center in Tel Hashomer, Israel. Using advertisements at each site, we recruited men age 30-65 with major depressive disorder incompletely responsive to a serotonergic antidepressant, and showing a total testosterone level ≤ 350 ng/dL.
Pre-assignment Details: At baseline, participants began a 1-week, single-blind placebo lead-in of one packet of placebo gel daily. Men exhibiting ≥ 50% improvement on either the Hamilton Depression Rating Scale (HAM-D) or Montgomery-Asberg Depression Rating Scale (MADRS) after placebo lead-in were withdrawn; all others were randomized to study medication.
Groups:
- Testosterone Gel: AndroGel, (1% testosterone transdermal gel), 2.5 g - 10 g daily
- Placebo Gel: Placebo gel identical in appearance to the testosterone gel
Period: Overall Study
Arm/Group | Testosterone Gel | Placebo Gel
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Testosterone Gel | Placebo Gel | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 50 | 100
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 50.6 (8.2) | 49.9 (7.1) | 50.3 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 50 | 50 | 100
Region of Enrollment [Number; unit: participants]
  United States | 29 | 24 | 53
  Israel | 21 | 26 | 47

OUTCOME MEASURES:

1. Secondary Outcome: Montgomery Asberg Depression Rating Scale (MADRS)
Description: The Montgomery Asberg Depression Rating Scale (MADRS) is a clinician-assessed scale that rates depressive symptoms on a scale from 0 (no depressive symptoms) to 60 (maximal depressive symptoms).
Time Frame: 9 weeks (1 week of placebo lead-in and 8 weeks of blinded medication treatment)
Population: All of the 100 randomized participants are included in the Last Observation Carried Forward (LOCF) analysis presented here online, which provides the mean and SD of this outcome measure for each study arm. Full details of all analyses are provided in the published paper presenting the results of the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Testosterone Gel | Placebo Gel
Number analyzed (Participants) | 50 | 50
units on a scale | 17.9 (9.0) | 19.9 (8.4)

2. Primary Outcome: 21-item Hamilton Depression Rating Scale Score (HAM-D)
Description: The HAM-D generates a score ranging from 0 (no depressive symptoms) to 64 (most severe depression).
Time Frame: 9 weeks (1-week placebo lead-in and 8 weeks of blinded medication treatment)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Testosterone Gel | Placebo Gel
Number analyzed (Participants) | 50 | 50
units on a scale | 13.5 (7.1) | 15.6 (6.2)
Statistical Analysis 1: Comparison: Testosterone Gel vs Placebo Gel; Our primary analysis of efficacy was a mixed effects linear regression analysis comparing the rate of change of score on the HAM-D during the blinded treatment phase between groups. Our model for the mean of the outcome variable included terms for treatment, time (modeled as a continuous variable), and treatment-by-time. The measure of effect was the treatment-by-time interaction, which can be interpreted as the difference in slope with respect to time, of the outcome measure; Test type: Superiority or Other; p = 0.71, mixed effects linear regression analysis — For a complete presentation of the above analysis, please see the published paper presenting the full results of this study

ADVERSE EVENTS:
Time Frame: Adverse events were assessed at all study visits throughout the eight-week blinded phase of the study.
Arm/Group | Testosterone Gel | Placebo Gel
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 3/50 | 0/50
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Testosterone Gel (N=50) | Placebo Gel (N=50)
headache (Nervous system disorders) | 3 (3) | 0 (0)

LIMITATIONS AND CAVEATS:
The small number of participants limited statistical power. Also, the study recruited "treatment-resistant" men, who are often poorly responsive. For a detailed discussion, see the published report of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No